CLINICAL TRIAL: NCT01752530
Title: A Study of the Efficacy of Computerized Cognitive Training on Cognitive Function, Symptoms and Functional Outcome in Children With ADHD.
Brief Title: Cognitive Training in Children With Attention Deficit/ Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Syddanmark (Other)
Responsible Party: Principal Investigator, Aida Bikic, psychologist, Ph.D. student, Region Syddanmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-20120096
Record Dates: First submitted 2012-12-10; First posted 2012-12-19 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: ADHD
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Cognitive Training; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer program C8 + treatment as usual (Experimental): Computer program C 8 + treatment as usual. Subjects in the intervention group will be playing a special computer program C8 for 40 min a day, 6 times a week for 8 weeks in addition to treatment as usual.
  Interventions: Other: Computer program C8; Other: Treatment as usual
- Treatment as usual (Other): Treatment as usual at the clinic
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Computer program C8 — Experimental: Computer program C8 + treatment as usual: Playing a special computer program C8 40 min a day for 6 days a week for 8 weeks.
  Other Names: C8; ADHD; Cognitive training
  Arms: Computer program C8 + treatment as usual
Other: Treatment as usual — Treatment as usual at the clinic
  Other Names: TAU

SUMMARY:
The purpose of this study is to determine the effect of computer program C8 on specific cognitive functions, symptoms and functional outcome compared to treatment as usual in children with ADHD. Furthermore, if the effect is sustained 12 and 24 weeks after training. In addition, it will be investigated, whether younger children benefit more from training than older children.

ELIGIBILITY:
Inclusion Criteria:

1. ADHD- diagnosis
2. age 6-13 years
3. Patient has access to computer og internet from home
4. Informed consent

Exclusion Criteria:

1. Comorbidity: conduct disorder, autism spectrum disorders, depression, or schizophrenia
2. Head trauma or neurological disease
3. Intelligence quotient (IQ) < 80
4. Motoric or perceptual handicap
5. Medical disease requiring treatment
6. No informed consent

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cambridge Neuropsychological Test Automated Battery (CANTAB): Rapid Visual Information Processing probability of hit. | Assesment after the 8 week intervention

SECONDARY OUTCOMES:
Behavior Rating Inventory of Executive Functions (BRIEF) | After the 8 week intervention
ADHD-Rating scale | After the 8 week intervention
CANTAB: Attention Switching Task (AST) | After the 8 week intervention
Cambridge Neuropsychological Test Automated Battery (CANTAB): Rapid Visual Information Processing | After 8 weeks of intervention

OTHER OUTCOMES:
CANTAB: Match to sample: visual search. | After 8 weeks of intervention
CANTAB: Choice reaction time. | After 8 weeks of intervention
CANTAB: Stop Signal Task. | After 8 weeks of intervention
CANTAB: Spatial Working Memory | After the 8 weeks of intervention
CANTAB: Stockings of Cambridge. | After the 8 weeks of intervention
CANTAB: Paired Associates Learning. | After 8 weeks of intervention
Weis function scale | After 8 weeks of intervention
Behavior Rating Inventory of Executive Functions (BRIEF) | 12 weeks follow up
Behavior Rating Inventory of Executive Functions (BRIEF) | 24 week follow up
ADHD-Rating scale | 12 week follow up
ADHD-Rating scale | 24 week follow up
CANTAB: Attention Switching Task (AST) | 12 week follow up
CANTAB: Attention Switching Task (AST) | 24 week follow up
CANTAB: Match to sample: visual search. | 12 week follow up
CANTAB: Match to sample: visual search. | 24 week follow up
CANTAB: Choice reaction time. | 12 weeks follow up
CANTAB: Choice reaction time. | 24 week follow up
CANTAB: Stop Signal Task. | 12 weeks follow up
CANTAB: Stop Signal Task. | 24 week follow up
CANTAB: Spatial Working Memory | 12 week follow up
CANTAB: Spatial Working Memory | 24 week follow up
CANTAB: Stockings of Cambridge. | 12 weeks follow up
CANTAB: Stockings of Cambridge. | 24 weeks follow up
Weis function scale | 12 week follow up
Weis function scale | 24 week follow up

CONTACTS AND LOCATIONS:
Overall Officials: Aida Bikic, Ph.D, Principal Investigator — Child and Adolescent Mental Health Services; Søren Dalsgaard, MD, Ph.D., Study Chair — Department of Economics and Business - CIRRAU - Centre for Integrated Register-based Research, Aarhus University
Locations (3):
- Denmark (3):
  - Child and Adolescent Mental Health Services Aabenraa, Aabenraa
  - Child and Adolescent Mental Health Services Augustenborg, Augustenborg
  - Child and Adolescent Mental Health Services Kolding, Kolding

REFERENCES:
- [Derived] Bikic A, Leckman JF, Christensen TO, Bilenberg N, Dalsgaard S. Attention and executive functions computer training for attention-deficit/hyperactivity disorder (ADHD): results from a randomized, controlled trial. Eur Child Adolesc Psychiatry. 2018 Dec;27(12):1563-1574. doi: 10.1007/s00787-018-1151-y. Epub 2018 Apr 11. PMID 29644473
- [Derived] Bikic A, Leckman JF, Lindschou J, Christensen TO, Dalsgaard S. Cognitive computer training in children with attention deficit hyperactivity disorder (ADHD) versus no intervention: study protocol for a randomized controlled trial. Trials. 2015 Oct 24;16:480. doi: 10.1186/s13063-015-0975-8. PMID 26499057